CLINICAL TRIAL: NCT04040868
Title: Safety and Accuracy of Robot-assisted Versus Fluoroscopy-assisted Screw Insertion in Spinal Surgery: a Prospective Multicenter Randomized Controlled Trial
Brief Title: Accuracy Study of Robot-assisted Screw Insertion in Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Wei Tian, President of Beijing Jishuitan Hospital, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JST-201903
Record Dates: First submitted 2019-04-10; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: the Robot-assisted Technique

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robot-assisted technique (Other)
  Interventions: Device: the TiRobot system
- conventional fluoroscopy-assisted technique (Other)
  Interventions: Device: Freehand

INTERVENTIONS:
Device: the TiRobot system — The TiRobot system (TINAVI Medical Technologies Co. Ltd.) is a multi-indication orthopedic surgical robot that can be used in spinal, pelvic, and limb surgeries performed via an open or a minimally invasive approach
  Arms: robot-assisted technique
Device: Freehand — conventional fluoroscopy-assisted
  Arms: conventional fluoroscopy-assisted technique

SUMMARY:
The investigators present the design of a randomized trial to compare the accuracy and safety of screw insertion using the robot-assisted technique versus the conventional fluoroscopy-assisted technique in spine surgery at multicenter. The accuracy and safety of screw insertion are measured by deviation of guide pin placement position, deviation of screw placement position, and intraoperative or postoperative complications. Secondary outcome parameters such as radiation exposure, postoperative recovery, duration of surgery, length of hospital stay and economic appraisal were also evaluated and compared between treatment groups.

DETAILED DESCRIPTION:
In spinal surgery, the accurate placement of implants is the key to ensure the success of the surgery, to achieve the safety and clinical requirements of internal fixation. Robot-assisted technology has become an effective means to improve the accuracy of implants with higher accuracy, free from fatigue and equivalent repetitive operation. The investigators present the design of a randomized trial to compare the accuracy and safety of screw insertion using the robot-assisted technique versus the conventional fluoroscopy-assisted technique in spine surgery at multicenter.

500 participants per group (1000 participants in total) are being recruited after diagnosis and before treatment through multi-hospital system and randomised to 1) robot-assisted technique or 2) conventional fluoroscopy-assisted technique in spine surgery. Outcomes are being measured pre-operatively, during- surgery and at 3, 6, 12 months post-surgery. The accuracy and safety of screw insertion are measured by deviation of guide pin placement position, deviation of screw placement position, and intraoperative or postoperative complications. Secondary outcome parameters such as radiation exposure, postoperative recovery, duration of surgery, length of hospital stay and economic appraisal were also evaluated and compared between treatment groups.

The study is addressing key questions of importance by evaluating the TiRobot-assisted technique versus the conventional fluoroscopy-assisted technique in spine surgery at multicenter. Outputs include evidence to facilitate more effective and safe decision making about surgical treatment for spine.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or above, gender not limited;
* patients eligible for surgery;
* the patient signed the informed consent and agreed to participate in this study.

Exclusion Criteria:

* patients with severe osteoporosis;
* patients with old fractures;
* patients with developmental deformity of the vertebral body with screw placement;
* patients complicated with severe systemic diseases;
* patients with coagulation dysfunction;
* patients deemed unsuitable for the test by the clinical institution.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Deviation of guide pin placement position | during operation
  After completing guide pin placement preparation, do the C arm scan, obtain 3-D scanning image, plan on the image, position by the robot, finish the needle placement and obtain 3-D scanning image again. Fusion two groups of the image, measure the distance between the entry and exit points of the guide pin and the surgical planning, calculate the insertion deviation, and evaluate the insertion accuracy of the guide pin.
  Insertion deviation = (Input offset distance + Output offset distance) / 2, the unit is mm.
  If more than one guide pin is needed for the operation, the deviation of the insertion shall be calculated separately and the average shall be taken.
Time of guide pin adjustion | during operation
  After the guide pin is placed, when the position deviation needs to be adjusted, the time consumed by adjusting the guide pin.
Deviation of screw placement position | during operation
  Postoperative screw placement position deviation was measured.
  The position of spinal screws was evaluated by postoperative imaging. Standard for classification of spinal screw placement :
  Excellent：The screw was completely in the pedicle and did not penetrate the cortex.
  Good: The screw cortical perforation < 2mm, or less than 50% of the screw diameter.
  Bad： The screw cortical perforation > 2mm, or more than 50% of the screw diameter.
Time of screw adjustion | during operation
  After the screw is placed, when the position deviation needs to be adjusted, the time consumed by adjusting the screw.
Intraoperative Complications | After operation up to 4 weeks
  Intraoperative complications, including but not limited to: positioning complications (blindness, nerve injury, skin breakdown), acute spinal cord injury, vascular Injury(vertebral injury, aorto-iliac injury), cardiovascular events, pulmonary complications, acute kidney injury.
Postoperative Complications | The time was within 1 year after the operation.
  Postoperative complications，including but not limited to: cardiovascular events, pulmonary complications, acute kidney injury, ileus, coagulopathy and wound infection. The time was within 1 year after the operation.

SECONDARY OUTCOMES:
Duration of surgery | during operation
  Duration of surgery refers to the time from the end of anesthesia to the end of the operation. In addition to the total operation time, the time before the screw placement, the time used for the screw placement, the time used for intraoperative decompression or reduction (if any) and the time used for install connecting rod were separately counted.
Radiation exposure | during operation
  Measure and calculate the radiation exposure to the patients and clinicians.
Visual analogue scale (VAS) score 24 hours before surgery | 24 hours before surgery
  Patients' pain information was evaluated by VAS score. The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Visual analogue scale (VAS) score 24 hours after surgery | 24 hours after surgery
  Patients' pain information was evaluated by VAS score. The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Visual analogue scale (VAS) score 3 months after surgery | 3 months after surgery
  Patients' pain information was evaluated by VAS score. The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Visual analogue scale (VAS) score 6 months after surgery | 6 months after surgery
  Patients' pain information was evaluated by VAS score. The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Visual analogue scale (VAS) score 1 year after surgery | 1 year after surgery
  Patients' pain information was evaluated by VAS score. The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
JOA score 24 hours before surgery | 24 hours before surgery
  For patients with cervical vertebra diseases, a 17-point cervical JOA score was used to evaluate the spinal cord function. For patients with lumbar vertebral disease, a 29-point lumbar JOA score was used to evaluate spinal cord function. JOA scores of the patients were collected before surgery, after surgery, and 3 months, 6 months and 1 year postoperatively.
JOA score 24 hours after surgery | 24 hours after surgery
  For patients with cervical vertebra diseases, a 17-point cervical JOA score was used to evaluate the spinal cord function. For patients with lumbar vertebral disease, a 29-point lumbar JOA score was used to evaluate spinal cord function. JOA scores of the patients were collected before surgery, after surgery, and 3 months, 6 months and 1 year postoperatively.
JOA score 3 months after surgery | 3 months after surgery
  For patients with cervical vertebra diseases, a 17-point cervical JOA score was used to evaluate the spinal cord function. For patients with lumbar vertebral disease, a 29-point lumbar JOA score was used to evaluate spinal cord function. JOA scores of the patients were collected before surgery, after surgery, and 3 months, 6 months and 1 year postoperatively.
JOA score 6 months after surgery | 6 months after surgery
  For patients with cervical vertebra diseases, a 17-point cervical JOA score was used to evaluate the spinal cord function. For patients with lumbar vertebral disease, a 29-point lumbar JOA score was used to evaluate spinal cord function. JOA scores of the patients were collected before surgery, after surgery, and 3 months, 6 months and 1 year postoperatively.
JOA score 1 year after surgery | 1 year after surgery
  For patients with cervical vertebra diseases, a 17-point cervical JOA score was used to evaluate the spinal cord function. For patients with lumbar vertebral disease, a 29-point lumbar JOA score was used to evaluate spinal cord function. JOA scores of the patients were collected before surgery, after surgery, and 3 months, 6 months and 1 year postoperatively.
NDI score 24 hours before surgery | 24 hours before surgery
  For patients with cervical vertebra diseases, NDI score was used to evaluate cervical spine dysfunction index. Total score from 0 (no disability) to 50 (complete disability).
NDI score 24 hours after surgery | 24 hours after surgery
  For patients with cervical vertebra diseases, NDI score was used to evaluate cervical spine dysfunction index. Total score from 0 (no disability) to 50 (complete disability).
NDI score 3 months after surgery | 3 months after surgery
  For patients with cervical vertebra diseases, NDI score was used to evaluate cervical spine dysfunction index. Total score from 0 (no disability) to 50 (complete disability).
NDI score 6 months after surgery | 6 months after surgery
  For patients with cervical vertebra diseases, NDI score was used to evaluate cervical spine dysfunction index. Total score from 0 (no disability) to 50 (complete disability).
NDI score 1 year after surgery | 1 year after surgery
  For patients with cervical vertebra diseases, NDI score was used to evaluate cervical spine dysfunction index. Total score from 0 (no disability) to 50 (complete disability).
ODI score 24 hours before surgery | 24 hours before surgery
  For patients with lumbar vertebra diseases, ODI score was used to evaluate the lumbago related score. The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain.
  0% -20%: Minimal disability 21%-40%: Moderate Disability 41%-60%: Severe Disability 61%-80%: Crippling back pain 81%-100%: These patients are either bed-bound or have an exaggeration of their symptoms.
ODI score 24 hours after surgery | 24 hours after surgery
  For patients with lumbar vertebra diseases, ODI score was used to evaluate the lumbago related score. The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain.
  0% -20%: Minimal disability 21%-40%: Moderate Disability 41%-60%: Severe Disability 61%-80%: Crippling back pain 81%-100%: These patients are either bed-bound or have an exaggeration of their symptoms.
Health related quality of life 3 months after surgery | 3 months after surgery
  Health related quality of life is being assessed with the SF-36 that is the most widely used QOL measure in the world with norms for the Australian general population available. The SF-36 contains a mental health and physical health summary scale suitable to measure the impact of the intervention on patients' wellbeing.
Health related quality of life 6 months after surgery | 6 months after surgery
  Health related quality of life is being assessed with the SF-36 that is the most widely used QOL measure in the world with norms for the Australian general population available. The SF-36 contains a mental health and physical health summary scale suitable to measure the impact of the intervention on patients' wellbeing.
Health related quality of life 1 year after surgery | 1 year after surgery
  Health related quality of life is being assessed with the SF-36 that is the most widely used QOL measure in the world with norms for the Australian general population available. The SF-36 contains a mental health and physical health summary scale suitable to measure the impact of the intervention on patients' wellbeing.
Economic appraisal | The time was within 1 year after the operation.
  Costs for each arm of the trial will be analysed by components of the intervention pathway (e.g. pre-consultation, work-up, theatre, post-treatment, follow-up, management/coordination, side-effects, etc.); by expenditure category (e.g. capital, staff, consumables, overheads, other); and by incidence (i.e. who bears the costs). The cost component of the economic appraisal will thus assess the cost drivers from a range of perspectives for both intervention approaches. Downstream costs and potential cost offsets incurred beyond the randomized trial data collection period will be modelled from the literature and expert opinion, with sources clearly documented.
length of hospital stay | Up to the 4 weeks
  Length of hospital stay refers to the time from the first day of hospitalization to the discharge after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Jishuitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan M, Fang Y, Zhang Q, Zhao J, Liu B, Tian W. A prospective cohort study of the accuracy and safety of robot-assisted minimally invasive spinal surgery. BMC Surg. 2022 Feb 11;22(1):47. doi: 10.1186/s12893-022-01503-4. PMID 35148734